CLINICAL TRIAL: NCT02390414
Title: The Myelodysplasia Transplantation-Associated Outcomes (MDS-TAO) Study
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Gregory A. Abel, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 11-056
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Results first posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Myelodysplastic Syndromes (MDS)
Keywords: Myelodysplastic syndromes (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gets HSCT: Patients with higher-risk myelodysplastic syndrome (MDS) aged 60-75 who are fit for HSCT and actually undergo HSCT.
- No HSCT: Patients with higher-risk myelodysplastic syndrome (MDS) aged 60-75 who are fit for HSCT but do not undergo HSCT.

SUMMARY:
The purpose of this observational study is to compare overall survival in older adults with myelodysplastic syndromes (MDS) who receive reduced intensity conditioning hematopoietic stem cell transplant (RIC HSCT) versus those who do not receive HSCT.

DETAILED DESCRIPTION:
MDS is a hematologic malignancy characterized by cytopenias, bone marrow failure, and a risk of transformation to acute myeloid leukemia (AML). HSCT is the only curative therapy for MDS. Despite its increasing use among older patients (age greater than 60), more data are needed to assess outcomes of HSCT in older adults compared to other therapies.

In this observational study, patients with MDS presenting at the study institutions are screened for disease characteristics that indicate that they are potentially appropriate for HSCT (both high-risk disease and fit for the procedure). Patients who meet inclusion and exclusion criteria and agree to participate in the study are entered into a clinical database and followed for overall survival. Patients also complete quality of life (QoL) assessments at enrollment and two years afterward, with the goal of investigating potential relationships between QoL and MDS treatment (HSCT vs. non-HSCT strategies).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of:

  * Primary or secondary MDS using the World Health Organization (WHO) 2008 classification:

    * Refractory cytopenia with unilineage dysplasia

      * Refractory Anemia (RA)
      * Refractory Neutropenia (RN)
      * Refractory Thrombocytopenia (RT)
    * Refractory Anemia with Ring Sideroblasts (RARS)
    * Refractory Cytopenia with Multilineage Dysplasia (RCMD)
    * Refractory Anemia with Excess Blasts-1 (RAEB-1)
    * Refractory Anemia with Excess Blasts-2 (RAEB-2)
    * MDS with isolated del (5q)
    * MDS-Unclassified (MDS-U)
  * Another of the following related disorders:

    * Chronic Myelomonocytic leukemia (CMML)
    * Myelodysplastic/myeloproliferative neoplasm, unclassifiable (MDS/MPD-U)
* Age 60 to 75 years
* Any of the following (high-risk characteristics):

  * Intermediate-2 or High-Risk on International Prognostic Scoring System (IPSS)
  * Secondary MDS (any karyotype)
  * Documented non-IPSS intermediate- or poor-prognosis karyotype including:

    * +8
    * t(11q23)
    * Rea 3q
    * +19
    * 3 or greater abnormalities
    * del(7q)
    * -5
    * t(5q)
  * Documented significant cytopenia for at least four months prior to enrollment, defined by the following criteria:

    * Red Blood Cell (RBC) Transfusion Dependence: four or more units of RBC transfusions within an eight-week period for symptomatic anemia with hemoglobin of ≤ 9.0 g/dL; OR
    * Severe Anemia: average of two or more hemoglobin values ≤ 8 g/dL within an eight-week period not influenced by RBC transfusions (i.e., must be seven days post transfusion); OR
    * Severe Thrombocytopenia: average of two or more platelet counts ≤ 50

      × 109/L within an eight-week period not influenced by platelet transfusions (i.e., must be at least three days post- transfusion) or a clinically significant hemorrhage requiring platelet transfusions within the prior four months; OR
    * Severe Neutropenia: average of two or more absolute neutrophil counts (ANC) ≤ 500 within an eight-week period, or a clinically significant infection requiring IV antibiotics in the setting of ANC ≤ 1000 within the prior four months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Adequate organ function to permit RIC HSCT as indicated by the following:

  * Serum bilirubin ≤ 2.5 mg/dL (except when Gilbert's syndrome or MDS-related hemolysis suspected).
  * Aspartate aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN).
  * Serum creatinine ≤ 2.0 mg/dL.
  * Seemingly sufficient baseline cardiac function to undergo HSCT (no echocardiogram required).
  * Seemingly sufficient baseline pulmonary function to undergo HSCT (no pulmonary function tests required).
  * Seemingly sufficient neuro-psychiatric function to undergo HSCT (no specific neuro-psychiatric evaluation required).
* Willingness to undergo human leukocyte antigen (HLA)-typing and consider subsequent HSCT.
* Willingness and ability to give informed consent.

Exclusion Criteria:

* Known baseline conversion to AML (eg, ≥ 20% peripheral or marrow blasts).
* Knowledge of potential donor status at study entry. Of note, knowledge of HLA status WITHOUT a related or unrelated search is allowed.
* History of prior malignancy within the past year, except for adequately-treated carcinoma in situ of uterine cervix, basal cell or squamous cell skin cancer.
* Any severe concurrent disease, infection, or comorbidity that, in the judgment of the principal investigator, would make the patient inappropriate for HSCT at the time of study entry.
* Psychiatric disorders including dementia that would preclude obtaining informed consent or the ability to participate in an ongoing research study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be 60 to 75 years old with a diagnosis of MDS or related disorder (eg, MDS/MPD or CMML) who have disease that is advanced enough to warrant RIC HSCT (defined by high-risk cytogenetics OR int-2 or high-risk on IPSS OR transfusion dependence as defined by WPSS) and who are physically fit enough to undergo RIC HSCT as assessed by pre-determined measures of organ function. Patients whose baseline donor status is known will be excluded; however, knowledge of HLA status is allowed as long as a donor search has not been performed.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Abel, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- See also: Fit older adults with advanced myelodysplastic syndromes: who is most likely to benefit from transplant? — https://doi.org/10.1038/s41375-020-01092-2

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gets HSCT | No HSCT
Started | 113 | 177
Completed | 113 | 177
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gets HSCT | No HSCT | Total
Number analyzed (Participants) | 113 | 177 | 290
Age, Continuous [Median (Full Range); unit: years] | 67 [60 to 75] | 70 [60 to 75] | 69 [60 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 60 | 100
  Male | 73 | 117 | 190
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 110 | 168 | 278
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Scale.
  0= Fully active, able to carry on all pre-disease performance without restriction. 1= Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. 2= Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. 3= Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  Participants
    0 | 37 | 53 | 90
    1 | 69 | 99 | 168
    2 | 7 | 24 | 31
    3 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: To prospectively compare the overall survival of patients in the HSCT group to that of patients in the non-HSCT group.
Time Frame: 3 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Gets HSCT | No HSCT
Number analyzed (Participants) | 113 | 177
Participants | 55 | 58

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed for 3 years
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Gets HSCT | No HSCT
All-Cause Mortality (participants affected / at risk) | 58/113 | 119/177
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT02390414/Prot_SAP_000.pdf